CLINICAL TRIAL: NCT04601064
Title: Peer Supported Collaborative Care to Increase Engagement in Mental Health and Substance Use Disorder Care in HIV Care Settings
Brief Title: Peer Supported Collaborative Care Mental Health and Substance Use Disorder Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00264580; R01DA052297 (NIH)
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections; Substance Use Disorders; Mental Health Disorder; Addiction; Opioid Use; Drug Use
Keywords: Collaborative Care; Peer Support
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders; Mental Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborate Care (CC) Model (Experimental): For patients randomized to the CC arm, in addition to the provider being alerted to the positive Mental Health and Substance Use Disorder screener, the patient will also be assigned to a peer case manager (P-CM). The P-CM will provide longitudinal care for the patient as part of their care management case load. The collaborative care support team will include the P-CM, a consultant addiction psychiatrist and the patient's HIV provider who will implement a stepped care program consisting of: 1) an initial assessment, determination of and implementation of an individualized care plan to provide; 2) psychosocial and medication adherence support; 3) evidence-based brief intervention incorporating motivational interviewing informed strategies; 4) measurement-based care for Mental Health and Substance Use Disorder provided directly by the HIV primary care provider or in collaboration with specialty Mental Health and Substance Use Disorder services.
  Interventions: Behavioral: Collaborative Care Model
- Usual Care (UC) (No Intervention): For patients randomized to the UC referral arm, the patient's HIV provider will receive an electronic alert of the patient's positive screen for a Mental Health and Substance Use Disorder. The patient will not be contacted by the P-CM. The provider, at their discretion, will initiate referral to the psychiatry service available onsite. For patients with Substance Use Disorder, providers refer to the in-clinic Substance Use Disorder treatment program that is managed by a nurse practitioner with Substance Use Disorder care experience. Once referred, the patient is seen by the nurse practitioner (separate from the HIV provider) who manages prescription of and assessment of adherence to buprenorphine, including monitoring of urine toxicology results with support from an addiction counselor. The Bartlett Clinic runs 2 substance use groups weekly and has processes for referral to a higher level of Substance Use Disorder care at offsite Substance Use Disorder treatment programs.

INTERVENTIONS:
Behavioral: Collaborative Care Model — Collaborative care (CC) is an evidence-based model of integrated mental health and substance use disorder care endorsed by the American Psychiatric Association for the integration of mental health and substance use disorder care into primary care settings. CC includes the following components: 1) A collaborative care team of multidisciplinary health care providers consisting of the primary physician, a care manager and a consulting psychiatrist, providing care in a coordinated fashion; 2) A population focus with the team working together to provide care and continuously measure and track health outcomes of a defined population of patients; 3) A measurement-guided approach with systematic use of disease specific patient reported outcome measures, such as symptom rating scales like the PHQ-9 to drive clinical decision making; and 4) Evidence-based practices with the team adapting scientifically proven treatments within an individual clinical context to achieve improved health outcomes.
  Arms: Collaborate Care (CC) Model

SUMMARY:
This is a research study to assess the effectiveness of a peer-led collaborative care model for integrating treatment for substance use and or mental health disorders into HIV care settings.

Depending on whether or not participants enroll in this study, participants will be assigned randomly (by chance, like drawing a number from a hat) to one of two groups. In group 1, participants would receive usual clinical care. In group 2, participants would work with a peer-case manager who would help support participants to engage in substance use or mental health disorder care. Regardless of the group participants are in, participants will fill out a survey when first enrolled in the study, and then again 12 months later.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18-99 years old
* accessing HIV care at the Bartlett HIV clinic
* Screened positive for a Mental health disorder or substance use disorder based on a computerized self-administered screen with Patient Health Questionnaire (PHQ-9)(score>10), General Anxiety Disorder (GAD-7) (score>10), National Institute on Drug Abuse Drug Use Screening Tool: 3 Question Quick Screen (Response of "Yes" to one or more heavy drinking days or "Yes" to use of illegal drugs or prescription drugs for non-medical reasons.
* Does not currently have a Mental Health or Substance Use Disorder treatment provider and or not receiving any current treatment (psychotherapy or pharmacotherapy) for Mental Health or Substance Use Disorder.
* English speaking

Exclusion Criteria:

• Individuals lacking the capacity to consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
The Number of Participants with HIV Virologic Suppression | Within a 3 month window of the 12 month follow-up (i.e. 3 months before or after the 12 month follow up)
  This is defined as a viral load < 200 copies/ml

SECONDARY OUTCOMES:
Number of Participants with Retention in HIV Care | Within 12 months of patient entrance into the study
  At least 2 medical visit dates, specifically for HIV care, that are at least 90 days apart
Number of Participants Who Obtain Treatment for Mental Health and Substance Use Disorder | Within 12 month of patient entrance into the study
  Receipt of evidence-based treatment for Mental Health and Substance Use Disorder, including medication and brief psychotherapy
Number of Participants with Change in Severity of Mental Health and Substance Use Disorder | Changes from baseline to 12 month follow up
  The following changes in Mental Health and Substance Use Disorder outcomes from baseline to 12 month follow up: Depression- 50% reduction in PHQ 9, Anxiety- 50% reduction in GAD 7, Bipolar Disorder- 50% reduction in Altman Mania Scores, PTSD- 50% reduction in PTSD Checklist 5, and Substance Use Disorder- 50% reduction in severity of dependence scale score

CONTACTS AND LOCATIONS:
Overall Officials: Oluwaseun Falade-Nwulia, MBBS, MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vagenas P, Azar MM, Copenhaver MM, Springer SA, Molina PE, Altice FL. The Impact of Alcohol Use and Related Disorders on the HIV Continuum of Care: a Systematic Review : Alcohol and the HIV Continuum of Care. Curr HIV/AIDS Rep. 2015 Dec;12(4):421-36. doi: 10.1007/s11904-015-0285-5. PMID 26412084
- [Background] Chander G, Himelhoch S, Moore RD. Substance abuse and psychiatric disorders in HIV-positive patients: epidemiology and impact on antiretroviral therapy. Drugs. 2006;66(6):769-89. doi: 10.2165/00003495-200666060-00004. PMID 16706551
- [Background] Azar MM, Springer SA, Meyer JP, Altice FL. A systematic review of the impact of alcohol use disorders on HIV treatment outcomes, adherence to antiretroviral therapy and health care utilization. Drug Alcohol Depend. 2010 Dec 1;112(3):178-93. doi: 10.1016/j.drugalcdep.2010.06.014. Epub 2010 Aug 11. PMID 20705402
- [Background] Rooks-Peck CR, Adegbite AH, Wichser ME, Ramshaw R, Mullins MM, Higa D, Sipe TA; Prevention Research Synthesis Project. Mental health and retention in HIV care: A systematic review and meta-analysis. Health Psychol. 2018 Jun;37(6):574-585. doi: 10.1037/hea0000606. PMID 29781655
- [Background] Chander G, Himelhoch S, Fleishman JA, Hellinger J, Gaist P, Moore RD, Gebo KA. HAART receipt and viral suppression among HIV-infected patients with co-occurring mental illness and illicit drug use. AIDS Care. 2009 May;21(5):655-63. doi: 10.1080/09540120802459762. PMID 19444675
- [Background] Sam TS, Hutton HE, Lau B, McCaul ME, Keruly J, Moore R, Chander G. Antiretroviral Therapy Use, Medication Adherence, and Viral Suppression Among PLWHA with Panic Symptoms. AIDS Behav. 2015 Nov;19(11):2049-56. doi: 10.1007/s10461-015-1064-4. PMID 25903506
- [Background] Monroe AK, Lau B, Mugavero MJ, Mathews WC, Mayer KH, Napravnik S, Hutton HE, Kim HS, Jabour S, Moore RD, McCaul ME, Christopoulos KA, Crane HC, Chander G. Heavy Alcohol Use Is Associated With Worse Retention in HIV Care. J Acquir Immune Defic Syndr. 2016 Dec 1;73(4):419-425. doi: 10.1097/QAI.0000000000001083. PMID 27243904
- [Background] Chander G, Lau B, Moore RD. Hazardous alcohol use: a risk factor for non-adherence and lack of suppression in HIV infection. J Acquir Immune Defic Syndr. 2006 Dec 1;43(4):411-7. doi: 10.1097/01.qai.0000243121.44659.a4. PMID 17099312
- [Background] Falade-Nwulia O, Sutcliffe CG, Mehta SH, Moon J, Chander G, Keruly J, Katzianer J, Thomas DL, Moore RD, Sulkowski MS. Hepatitis C Elimination in People With HIV Is Contingent on Closing Gaps in the HIV Continuum. Open Forum Infect Dis. 2019 Sep 30;6(10):ofz426. doi: 10.1093/ofid/ofz426. eCollection 2019 Oct. PMID 31667200
- [Background] Westergaard RP, Hess T, Astemborski J, Mehta SH, Kirk GD. Longitudinal changes in engagement in care and viral suppression for HIV-infected injection drug users. AIDS. 2013 Oct 23;27(16):2559-66. doi: 10.1097/QAD.0b013e328363bff2. PMID 23770493
- [Background] Campo RE, Alvarez D, Santos G, Latorre J. Antiretroviral treatment considerations in Latino patients. AIDS Patient Care STDS. 2005 Jun;19(6):366-74. doi: 10.1089/apc.2005.19.366. PMID 15989432
- [Background] Giordano TP, Visnegarwala F, White AC Jr, Troisi CL, Frankowski RF, Hartman CM, Grimes RM. Patients referred to an urban HIV clinic frequently fail to establish care: factors predicting failure. AIDS Care. 2005 Aug;17(6):773-83. doi: 10.1080/09540120412331336652. PMID 16036264
- [Background] Lucas GM, Chaudhry A, Hsu J, Woodson T, Lau B, Olsen Y, Keruly JC, Fiellin DA, Finkelstein R, Barditch-Crovo P, Cook K, Moore RD. Clinic-based treatment of opioid-dependent HIV-infected patients versus referral to an opioid treatment program: A randomized trial. Ann Intern Med. 2010 Jun 1;152(11):704-11. doi: 10.7326/0003-4819-152-11-201006010-00003. PMID 20513828
- [Background] Low AJ, Mburu G, Welton NJ, May MT, Davies CF, French C, Turner KM, Looker KJ, Christensen H, McLean S, Rhodes T, Platt L, Hickman M, Guise A, Vickerman P. Impact of Opioid Substitution Therapy on Antiretroviral Therapy Outcomes: A Systematic Review and Meta-Analysis. Clin Infect Dis. 2016 Oct 15;63(8):1094-1104. doi: 10.1093/cid/ciw416. Epub 2016 Jun 25. PMID 27343545
- [Background] Sherer R, Stieglitz K, Narra J, Jasek J, Green L, Moore B, Shott S, Cohen M. HIV multidisciplinary teams work: support services improve access to and retention in HIV primary care. AIDS Care. 2002 Aug;14 Suppl 1:S31-44. doi: 10.1080/09540120220149975. PMID 12204140
- [Background] Saag LA, Tamhane AR, Batey DS, Mugavero MJ, Eaton EF. Mental health service utilization is associated with retention in care among persons living with HIV at a university-affiliated HIV clinic. AIDS Res Ther. 2018 Jan 16;15(1):1. doi: 10.1186/s12981-018-0188-9. PMID 29338735
- [Background] Ashman JJ, Conviser R, Pounds MB. Associations between HIV-positive individuals' receipt of ancillary services and medical care receipt and retention. AIDS Care. 2002 Aug;14 Suppl 1:S109-18. doi: 10.1080/09540120220149993a. PMID 12204145
- [Background] DeGroote NP, Korhonen LC, Shouse RL, Valleroy LA, Bradley H. Unmet Needs for Ancillary Services Among Men Who Have Sex with Men and Who Are Receiving HIV Medical Care - United States, 2013-2014. MMWR Morb Mortal Wkly Rep. 2016 Sep 23;65(37):1004-1007. doi: 10.15585/mmwr.mm6537a4. PMID 27657489
- [Background] Korhonen LC, DeGroote NP, Shouse RL, Valleroy LA, Prejean J, Bradley H. Unmet Needs for Ancillary Services Among Hispanics/Latinos Receiving HIV Medical Care - United States, 2013-2014. MMWR Morb Mortal Wkly Rep. 2016 Oct 14;65(40):1104-1107. doi: 10.15585/mmwr.mm6540a3. PMID 27736837
- [Background] Korthuis PT, Josephs JS, Fleishman JA, Hellinger J, Himelhoch S, Chander G, Morse EB, Gebo KA; HIV Research Network. Substance abuse treatment in human immunodeficiency virus: the role of patient-provider discussions. J Subst Abuse Treat. 2008 Oct;35(3):294-303. doi: 10.1016/j.jsat.2007.11.005. Epub 2008 Mar 7. PMID 18329222
- [Background] Oldfield BJ, Munoz N, McGovern MP, Funaro M, Villanueva M, Tetrault JM, Edelman EJ. Integration of care for HIV and opioid use disorder. AIDS. 2019 Apr 1;33(5):873-884. doi: 10.1097/QAD.0000000000002125. PMID 30882491
- [Background] Kaaya S, Eustache E, Lapidos-Salaiz I, Musisi S, Psaros C, Wissow L. Grand challenges: Improving HIV treatment outcomes by integrating interventions for co-morbid mental illness. PLoS Med. 2013;10(5):e1001447. doi: 10.1371/journal.pmed.1001447. Epub 2013 May 21. PMID 23700389
- [Background] Archer J, Bower P, Gilbody S, Lovell K, Richards D, Gask L, Dickens C, Coventry P. Collaborative care for depression and anxiety problems. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD006525. doi: 10.1002/14651858.CD006525.pub2. PMID 23076925
- [Background] Watkins KE, Ober AJ, Lamp K, Lind M, Setodji C, Osilla KC, Hunter SB, McCullough CM, Becker K, Iyiewuare PO, Diamant A, Heinzerling K, Pincus HA. Collaborative Care for Opioid and Alcohol Use Disorders in Primary Care: The SUMMIT Randomized Clinical Trial. JAMA Intern Med. 2017 Oct 1;177(10):1480-1488. doi: 10.1001/jamainternmed.2017.3947. PMID 28846769
- [Background] Pyne JM, Fortney JC, Curran GM, Tripathi S, Atkinson JH, Kilbourne AM, Hagedorn HJ, Rimland D, Rodriguez-Barradas MC, Monson T, Bottonari KA, Asch SM, Gifford AL. Effectiveness of collaborative care for depression in human immunodeficiency virus clinics. Arch Intern Med. 2011 Jan 10;171(1):23-31. doi: 10.1001/archinternmed.2010.395. PMID 21220657